CLINICAL TRIAL: NCT04599010
Title: Pilot Randomized Controlled Trial Comparing FFM-indexed Feeding vs. Standard Feeding in LGA Infants With Oral Feeding Difficulty and Disproportionate Body Composition.
Brief Title: Role of Body Composition in Large for Gestational Age Infants (LGA) With Oral Feeding Difficulty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Sreekanth Viswanathan, Attending Neonatologist, Professor of Pediatrics, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 871760
Record Dates: First submitted 2020-10-14; First posted 2020-10-22 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Body Composition; Feeding; Difficult, Newborn; Nutrition Disorder, Infant
MeSH Terms: conditions — Infant Nutrition Disorders | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: The sample size for this pilot study will be 40 with 20 infants randomized into each arm.
Who Masked: Outcomes Assessor
Masking Description: The data analyzer will be masked to the allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FFM-indexed feeding (Active Comparator): In FFM-indexed feeding, there will be a permissive feeding volume restriction to 150 ± 10 mL/kg (FFM)/day without increasing the milk calorie density or changing the type of formula milk for 2 weeks in the intervention group
  Interventions: Other: Dietary intervention
- Standard feeding (Active Comparator): The standard feeding approach will include an oral feeding volume goal of 150 ± 10 mL/kg/day during the 2-week study period
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — energy-restricted diet appropriate for resting metabolic rate using FFM as proxy

SUMMARY:
Large for Gestational Age (LGA) infants have excess fat-mass (FM) proportion secondary to prolonged in utero exposure to an energy-rich environment. Our preliminary data suggest that excess FM proportion can be associated with oral feeding delay and a potentially modifiable therapeutic target to improve oral feeding outcomes. The objective of this study is to determine the impact of a short-term Fat-free mass (FFM)-indexed feeding on the oral intake volumes in LGA infants with oral feeding difficulties.

DETAILED DESCRIPTION:
Eligible subjects will be randomized to an innovative FFM-indexed feeding or the standard feeding for up to 2 weeks. The essential component of the FFM-indexed feeding will be the difference in milk prescription dosing that we propose to set the feeding volume to index FFM rather than total mass. In FFM-indexed feeding, there will be a permissive feeding volume restriction to 150 ± 10 mL/kg (FFM)/day without increasing the milk calorie density or changing the type of formula milk, whereas the standard feeding will include a feeding volume goal of 150 ± 10 mL/kg (body weight)/day. Infants will receive either breast milk or formula feedings per the standard feeding protocols. Body composition (PEAPOD system) and appetite-regulating hormones (ARH) levels of enrolled infants will be assessed at baseline (test-1) and at the end 2-week study intervention period (test-2). Subjects will be followed for clinical and growth outcomes until neonatal intensive care unit (NICU) discharge and through 6 months of age. Growth will be followed through 6 months of age by retrieving anthropometric measurement records from pediatricians at well-child visits (2-, 4-, 6- and 6-month visits). Parents will be called at these time points to obtain a history of any further feeding difficulties.

ELIGIBILITY:
Inclusion Criteria:

* LGA infants with oral feeding difficulty born at ≥ 35 weeks gestation, with FM z-score > +1.0 in body composition measurement

Exclusion Criteria:

* Infants on any respiratory support, Infants on enteral feeding duration > 60 minutes due to hypoglycemia concerns, videofluoroscopic swallow study (VFSS) demonstrating unsafe swallowing function, GI surgical conditions, significant neurological morbidities, and major congenital, genetic syndromes/anomalies

Ages: 1 Week to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Time from study entry to independent oral feeding | Before or at NICU-discharge
  full oral feeding defined as 120 ml/kg/d without tube feeding for 2 consecutive days

SECONDARY OUTCOMES:
oral feeding volume at NICU discharge | before 3 months
  oral feeding volume (mL/kg/day) at discharge
NICU Feeding related length of stay (LOS) | before 3 months
  Days from first oral feeding to independent oral feeding
Gastrostomy rates | through study completion, an average of 1 year
  Percentage of infants with gastrostomy placement
ARH levels | 2 weeks
  Directional changes in ARH pre-post intervention
Oral feeding success rate | Before 3 months
  Independent oral feeding at NICU discharge
Body composition change in FM and FFM | 2 weeks
  Directional changes in FM and FFM pre-post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sreekanth Viswanathan, MD, Principal Investigator — Nemours Children's Clinic
Locations (2):
- United States (2):
  - Nemours Children's Hospital, Orlando, Florida
  - Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA)